CLINICAL TRIAL: NCT05104905
Title: A Phase I/II Open Label Single Centre Trial to Assess the Safety, Tolerability and Efficacy of Single Dose Neoadjuvant Anti-CLEVER-1 Antibody Bexmarilimab in Localised Renal Cell and Colon Carcinoma (Macrophage Antibody To Inhibit Immune Suppression in RENAl Cell and COLon Carcinomas)
Brief Title: A Phase I/II Open Label Single Centre Trial to Assess the Safety, Tolerability and Efficacy of Single Dose Neoadjuvant Anti-CLEVER-1 Antibody Bexmarilimab in Localised Renal Cell and Colon Carcinoma
Acronym: RENACOL
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Since no patients have been enrolled in RENACOL, and safety and tolerability data is rapidly accumulating in another ongoing study, sponsor considered that RENACOL study is no longer needed to assess the safety profile of bexmarilimab
Sponsor: Faron Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FP2CLI003; 2021-001030-19 (EudraCT Number)
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Carcinoma, Renal Cell; Carcinoma Colon
MeSH Terms: conditions — Carcinoma, Renal Cell; Colonic Neoplasms | interventions — bexmarilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Renal cell intervention 1.0 mg/kg (Experimental)
  Interventions: Drug: bexmarilimab
- Renal cell intervention 3.0 mg/kg (Experimental)
  Interventions: Drug: bexmarilimab
- Renal cell intervention 10 mg/kg (Experimental)
  Interventions: Drug: bexmarilimab
- Renal cell Observation (No Intervention)
- Colon cancer intervention 1.0 mg/kg (Experimental)
  Interventions: Drug: bexmarilimab
- Colon cancer intervention 3.0 mg/kg (Experimental)
  Interventions: Drug: bexmarilimab
- Colon cancer intervention 10 mg/kg (Experimental)
  Interventions: Drug: bexmarilimab
- Colon cancer Observation (No Intervention)

INTERVENTIONS:
Drug: bexmarilimab — A single neoadjuvant dose will be administered prior to surgery.
  Arms: Colon cancer intervention 1.0 mg/kg; Colon cancer intervention 10 mg/kg; Colon cancer intervention 3.0 mg/kg; Renal cell intervention 1.0 mg/kg; Renal cell intervention 10 mg/kg; Renal cell intervention 3.0 mg/kg

SUMMARY:
Bexmarilimab treatment has demonstrated tolerable safety profile and anticancer efficacy in some subjects with advanced malignancies. This is the first study to investigate the effect of single neoadjuvant dose of anti-CLEVER-1 antibody bexmarilimab prior to radical surgery of renal cell and colon cancers. We expect that the single dose will demonstrate measurable effects on the tumour immunological microenvironment as well as systemic effects on subject´s immunological status and that this evidence may be used to guide future neoadjuvant studies. There will be a dose escalation to investigate the effect of different doses of bexmarilimab. In addition to subjects receiving single neoadjuvant dose of bexmarilimab, there will be an observational cohort without Investigational Medicinal Product (IMP) for either cancer. All patients participating in the study (whether in investigational or observational cohort) will attend each visit and are assessed for the same endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Ability and stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged > 18 years.
4. Adequate general health (ECOG 0 or 1) to undergo planned radical surgery for renal cell or colon cancer.
5. Adequate bone marrow, liver and kidney function defined as: Blood white blood cell ≥ lower limit of normal Blood neutrophil count ≥ 1x109/L Blood platelet count ≥ 100x109/L Blood haemoglobin ≥ 9.0 g/dL Creatinine clearance > 40 mL/min calculated by Cockcroft-Gault formula Aspartate Aminotransferase (AST) ≤ 3 X Upper Limit of Normal (ULN) Alanine Aminotransferase (ALT) ≤ 3 X ULN Bilirubin ≤ 1.5 X ULN Albumin ≥ 3.0 g/dL
6. Histologically confirmed clear cell renal cell cancer planned to be treated with surgery with curative intent (Renal cell cancer cohort). In renal cell observation cohort, histological confirmation not mandatory.

   or Histologically confirmed adenocarcinoma of the colon planned to be treated with surgery with curative intent (Colon cancer cohort).

   Additional inclusion criteria for subjects planned to have a single neoadjuvant dose of CLEVER-1 antibody bexmarilimab:
7. For females of reproductive potential: use of highly effective contraception* for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 12 weeks after the end of single neoadjuvant dose of bexmarilimab administration.
8. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner during study participation and for an additional 12 weeks after the administration of single neoadjuvant dose of bexmarilimab.

   * Women of childbearing potential i.e. not post-menopausal or surgically sterilised must use highly effective methods of contraception. For example, combined estrogen and progestogen hormonal contraception to inhibit ovulation; progestogen-only hormonal contraception to inhibit ovulation; intra-uterine device (IUD); intrauterine hormone-releasing system (IUS) or vasectomised partner to prevent pregnancy or abstain. Abstinence must be in line with the preferred and usual lifestyle of the subject. Periodic abstinence such as calendar, ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception during heterosexual activity for the duration of the trial and for at least 12 weeks following the study drug administration. In addition, barrier contraception (with or without spermicide) may be used but this should not be considered as an adequate form of contraception on its own.

Fertile men whose partners could be of childbearing potential should routinely use a condom for 12 weeks after the study drug administration. The partner, if not pregnant, should also use a reliable form of contraception such as the oral contraceptive pill or an IUD.

Exclusion Criteria:

1. Evidence of metastatic disease making subject not eligible for surgical resection, except for local nodal metastatic disease.
2. History of previous treatment for renal cell cancer (renal cell cancer cohorts) or colon cancer (colon cancer cohorts).
3. Less than 3 months since the last dose of any cancer therapy prior to consenting.
4. Less than 4 weeks since any major surgery.
5. Treatment with any investigational agent within 4 weeks before consenting.
6. History of another malignancy without curative treatment or suspicion of disease recurrence.
7. Evidence of severe or uncontrolled systemic diseases, congestive cardiac failure New York Heart Association (NYHA) class 2, Myocardial Infarction (MI) within 6 months or laboratory finding that in the view of the investigator makes it undesirable for the subject to participate in the trial.
8. Any medical condition that the Investigator considers significant to compromise the safety of the subject or that impairs the interpretation of IMP toxicity assessment.
9. Confirmed human immunodeficiency virus infection.
10. Confirmed hepatitis B or C virus infection.
11. Symptomatic cytomegalovirus infection.
12. Subjects with active autoimmune disorder (except type I diabetes, celiac disease, hypothyroidism requiring only hormone replacement, vitiligo, psoriasis, or alopecia).
13. The subject requires systemic corticosteroid or other immunosuppressive treatment.
14. Subjects with organ transplants.
15. Subjects in dialysis.
16. Use of Live (attenuated) vaccines for 30 days prior to the start of study treatment, during treatment, and until last visit.
17. Subject is unwilling or unable to comply with treatment and trial instructions.
18. Pregnancy or lactation.
19. Medical history of chronic ulcers, abnormal liver function or previous liver problems/diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Adverse Events ≥Grade 3 during the 28 days (4 weeks) following the single dose of bexmarilimab and surgical adverse events ≥Grade 3 during the 14days (2 weeks) following the surgery | 28 days and 14 days
  Adverse Events ≥Grade 3 according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 during the 28 days (4 weeks) following the single dose of bexmarilimab and surgical adverse events ≥Grade 3 according to the Clavien-Dindo classification occurring during the 14 days (2 weeks) following the surgery

SECONDARY OUTCOMES:
Adverse events until the follow-up visit on Day 84 | Day 84
Radiological response rate according to the response evaluation criteria in solid tumours (RECIST 1.1) (Day 13) | Day 13
Pathological response rate evaluated with Ryan tumour regression grade (Day 14), percentage of tumour cell necrosis | Day 14
Long-term clinical benefit measured by disease-free survival assessed at 1, 3 and 5 years | 1, 3, and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Boström, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland